CLINICAL TRIAL: NCT05987098
Title: Safety and Clinical Value of 18Fluorine-labeled BBPA PET/CT in Patients With Malignant Tumors
Brief Title: BBPA PET/CT in Patients With Malignant Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-BBPA PET/CT
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Malignant Tumors
Keywords: malignant tumors; BBPA-PET/CT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A single dose of BBPA will be intravenously injected and PET examination will carry out 30 minutes later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malignant Tumors (Experimental): BBPA in suspected malignant tumors. This arm investigates the metabolic characteristics of BBPA in suspected malignant tumor patients who consider for surgical operations. A single dose of 0.10 mCi/kg BBPA will be intravenously injected and PET examination will carry out 30 minutes later. Surgical operations, if recommended after multiple examination, will be carried out within 1 week after BBPA PET scan.
  Interventions: Diagnostic Test: BBPA PET examination

INTERVENTIONS:
Diagnostic Test: BBPA PET examination — A single dose of 0.10 mCi/kg BBPA will be intravenously injected and PET examination will carry out 30 minutes later.

SUMMARY:
This study is an open-labeled phase II diagnostic clinical trial to explore the safety and clinical value of BBPA-PET/CT in suspected malignant tumor patients. The investigation regarding the clinical value of BBPA concerning the metabolic characteristics of BBPA in suspected malignant tumors. Quantitative features will be extracted to analysis the PET images. For patient who took surgery after multiple examination, histopathology, molecular pathology and LAT-1 immunohistochemistry will also be obtained.

DETAILED DESCRIPTION:
In this study, we utilized BBPA, a novel boron amino acid, which replaces the carboxyl group of 4-boronate phenylalanine (BPA) with a boron trifluoride group (-BF3) (-COOH), as a diagnostic molecule for PET imaging of brain tumors, is also a highly efficient boron carrier for BNCT. Preclinical studies suggested [18F]BBPA to be a pan-cancer probe that transmembrane transported through large neutral amino acid transporter type-1 (LAT-1). However more studies and evidence are warranted to investigate the clinical value of BBPA PET imaging in human.

This study aim to observe the safety of BBPA, and investigate the diagnostic value of BBPA in the patient with suspected malignant tumors. Patients who meet the eligibility criteria are included in clinical trials after fully communicating the condition, explaining the benefits and risks of clinical trials, clarifying the patient's willingness to include the clinical trial, and signing informed consent. The cohort number, BBPA administrative dose, imaging protocols are decided based on the investigators' preliminary data. The diagnosis and post- examination treatment are based on the recommended guideline, combined with the subject's own situation for standardized diagnosis and treatment

ELIGIBILITY:
Inclusion Criteria:

* Have suspected diagnosis of brain tumors, based on clinical performance and imaging results.
* Meet the indications for PET examination, show a clear indication and no contraindications;
* Have a performance status of score ≥80 on KPS scale or score 0-1 points on ECOG scale, a relatively good general situation;
* Does not appear agonal stage, deep coma, over grade 2 major organ dysfunction (heart, lung, liver, kidney and other major organ include), acute or life-threatening status of infection;
* Be ≥ 18 years of age on day of signing informed consent.
* Be willing and able to understand the research content and provide written informed consent/assent for the trial.

Exclusion Criteria:

* Have a history of imaging agent allergies;
* Does not meet the PET-CT scan sedation requirements, or there are contraindications for PET-CT examination;
* Be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial;
* Unable to adhere strictly to protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
standardized uptake value (SUV) for BBPA | 1 week
  SUV reflects the uptake of PET tracers, and quantitative imaging features such as SUVmax, SUVmean, and visually assessed features will be measured in the evaluation of tumors.

SECONDARY OUTCOMES:
Adverse events | 1 week
  Adverse event within 1 week after BBPA injection will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenbin Ma, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No